CLINICAL TRIAL: NCT03973385
Title: Evaluation of Efficacy of Cryotherapy for Skin Anesthesia During Arterial Puncture for Blood Gas in Critically Ill Patients. SNOW Study
Brief Title: Evaluation of Efficacy of Cryotherapy for Skin Anesthesia During Arterial Puncture
Acronym: SNOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Jacq Gwenaelle, Investigator coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P17/04_SNOW; 2018-A00702-53 (Other: Registry ID: ID RCB)
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Cryotherapy Effect
Keywords: cryotherapy; vapocoolant spray; arterial puncture; intensive care unit
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryotherapy group (Experimental): cryotherapy by vapocoolant spray is applied on skin for 4 to 10 seconds ( or up to skin whitening) to 15 centimeters distance with sweeping action before ABG
  Interventions: Device: Cryotherapy
- control group (Placebo Comparator): water spray is applied on skin for 4 to 10 seconds to centimeters distance with sweeping action before ABG
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Cryotherapy — patients recieving cryotherapy for skin anesthesia for artérial blood gas

SUMMARY:
the purpose of this study is to evaluate the cryotherapy effect by vapocoolant spray to reducing pain during puncture for artérial blood gas

DETAILED DESCRIPTION:
Blood gas analysis by arterial puncture is the Gold Standard in the assessment of a patient's acidbase status and oxygenation. This procedure, which can be repeated depending on the clinical condition of patient, is however associated with a potentially painful experience for patients.

The known anesthetic properties of cold can be an interesting alternative to evaluate in the reduction of pain induced during arterial puncture for gas analysis in critically il patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age≥18 years) hospitalized in Intensive Care Unit
* Patient requiering arteriale puncture for ABG
* A négative score of CAM ICU scale
* Patient with a score to visual analog scale < or equal 30mm
* Securité sociale affiliated
* consentement

Exclusion Criteria:

* patient undergoing mechanical ventilation
* patient with arterial catheter
* patient with arterio veinius fistul
* patient receiving topical anesthesic at least 2 h before the puncture
* patient with cutaneous lesion (zone of puncture)
* Raynaud Syndrom
* cold sensibility
* Allen test negative
* pregnant
* legal guardianship

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pain during arterial puncture | immediately after puncture
  Pain will be assessed with the visual analog scale (numeric value go 0 to 100 millimeters and representing intensity of pain from "no pain" to "worst pain imaginable"(1)

SECONDARY OUTCOMES:
Ease to performing Arterial Blood Gas (ABG) sampling | immediately after puncture
  Ease to performing ABG sampling will be evaluated by i)the number of punctures necessary to obtain a sample of at least 1ml of arterial blood, ii) the delay between the first arterial puncture, and obtaining a sample.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaëlle Jacq, RN, Principal Investigator — CH Versailles
Locations (4):
- France (4):
  - Hopital Nord Franche-Comte, Belfort
  - Ch Versailles, Le Chesnay
  - CHU Saint LOUIS, Paris
  - Hopital Européèn Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: No